CLINICAL TRIAL: NCT01141413
Title: Comparison of Dosing and Costs Between Rheumatoid Arthritis Patients Treated With Remicade® Versus Orencia®
Brief Title: Dose Escalation With Remicade® and Orencia®
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-255
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Last update posted 2012-04-04 (Estimated); Status verified 2012-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RA patients using Remicade®
- RA patients using Orencia®

SUMMARY:
The purpose of this study is to describe infliximab and abatacept dosing patterns (i.e., dosing amount and frequency) and costs among a population of managed care enrollees with RA. This study will also identify changes in infliximab and abatacept dosing over time and the implication these changes may have on the costs of medication administration.

DETAILED DESCRIPTION:
This study will be conducted in two parts. The primary analysis is a longitudinal analysis, where patients' health care claims from a period during which the patient was continuously enrolled in the health plan will be used to evaluate the primary outcome (i.e., dose escalation). The second analysis will be cross-sectional, where patients' health care claims from a fixed period of time (i.e., 2008) will be used to examine health care cost.

The final enrollment for the longitudinal portion of the study was 2,001 (1,306 infliximab and 695 abatacept patients). Final enrollment for the cross-sectional portion was 3,450 (2,646 infliximab and 806 abatacept patients). There may be some overlap in these numbers.

ELIGIBILITY:
Inclusion Criteria:

* Commercial health plan enrollees with medical and pharmacy coverage
* At least 3 claims on separate days for infliximab (HCPCS J1745) or abatacept (HCPCS C9230, J0129, J3590) administration during the subject identification period
* The 3 initial claims for abatacept occurred within a 6-week period inclusive of the index date and the three initial claims for infliximab occur within a 9-week period inclusive of the index date
* Presence of a diagnosis of RA (ICD-9-CM 714.xx)
* Continuous enrollment during the baseline and follow-up periods
* At least 18 years of age or older on the index date

Exclusion Criteria:

* Prior exposure to the index medication during the baseline period
* Diagnosis of psoriasis (ICD-9-CM 696.1), psoriatic arthritis (696.0), ankylosing spondylitis (720.0), Crohn's disease (555.x), or ulcerative colitis (556.x) in any position at any time during the study period
* Exposure to alefacept (HCPCS J0215, C9211, C9212) or efalizumab (HCPCS S0162) at any time during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Commercial health plan members
Sampling Method: Non-Probability Sample
Enrollment: 5451 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Escalation in dosing amount or frequency | Throughout follow-up period (variable, between 6 weeks and 39 months)

SECONDARY OUTCOMES:
Switch/discontinuation of index therapy | Throughout follow-up period (variable, between 6 weeks and 39 months)
Number of infusions | Throughout follow-up period (variable, between 6 weeks and 39 months)
Average dose per infusion | Throughout follow-up period (variable, between 6 weeks and 39 months)
Frequency of infusions | Throughout follow-up period (variable, between 6 weeks and 39 months)
Average costs per infusion | Throughout follow-up period (variable, between 6 weeks and 39 months)
Health care resource utilization | Throughout follow-up period (variable, between 6 weeks and 39 months)
Health care costs | Throughout follow-up period (variable, between 6 weeks and 39 months)
Concurrent medication use | Throughout follow-up period (variable, between 6 weeks and 39 months)
Time to maximum dose | Throughout follow-up period (variable, between 6 weeks and 39 months)
Time to dose escalation | Throughout follow-up period (variable, between 6 weeks and 39 months)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: BMS Clinical Trials Disclosure — http://www.bms.com/clinical_trials/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx
- See also: For FDA Safety Alerts and Recalls refer to the following link: http://www.fda.gov/MEDWATCH/safety.htm — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm